CLINICAL TRIAL: NCT06900322
Title: Structured and Specialized Physical Therapy: Does it Make a Difference for Children With Congenital Zika Syndrome?
Brief Title: Impacts of a Physical Therapy Protocol on Motor Function in Children With Congenital Zika Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriela Lopes Gama (Other)
Responsible Party: Sponsor-Investigator, Gabriela Lopes Gama, PhD, Instituto de Pesquisa Professor Joaquim Amorim Neto
Organization: Instituto de Pesquisa Professor Joaquim Amorim Neto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.839.838
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Congenital Zika Syndrome
MeSH Terms: conditions — Zika Virus Infection | interventions — Physical Therapy Modalities; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: Experimental Group (stimuli and handling; physical therapy [PediaSuit])
- Control group (Active Comparator)
  Interventions: Other: control group (conventional physical therapy)

INTERVENTIONS:
Other: Experimental Group (stimuli and handling; physical therapy [PediaSuit]) — Participants underwent a one-hour daily protocol (5 times a week) of stimuli and handling based on the neuroevolutionary concept, and motor physical therapy with therapeutic garments (PediaSuit).
  During therapy based in PediaSuit protocol therapy suits were used to stimulate proprioception, muscle contraction, and postural stability.Traction bands were placed on the trunk to stimulate muscle control by stabilizing this area and the antigravity muscles.The ability exercise unit was also used to stimulate postural stability and muscle resistance, according to the functional ability of each child.
  Neuroevolutionary concept is a problem-solving approach focused on the treatment of functional impairments, postural alignment and movement.
  Therefore, Neuroevolutionary concept is an individualised approach aimed at improving functionality and, consequently, the quality of life of individuals with neurological deficits.
  Arms: Experimental group
Other: control group (conventional physical therapy) — Participants kept the therapeutic routine (conventional physical therapy).
  Arms: Control group

SUMMARY:
The study aims to evaluate the effects of a specialized physiotherapy protocol aimed at the motor function of children with Congenital Zika Virus Syndrome. First, participants' anthropometric parameters (weight and length) and motor functions were assessed. After that participant were splited in two groups: Experimental group that uunderwent a one-hour daily protocol (5 times a week) of stimuli and handling based on the neuroevolutionary concept, and motor physical therapy with therapeutic garments (PediaSuit). On the other hand, the control group (CG) kept the therapeutic routine (conventional physical therapy).

ELIGIBILITY:
Inclusion Criteria:

* Children with confirmed CZS diagnosis by RT-PCR or presumed by imaging findings (CT or MRI [or both]), and according to the Center for Disease Control and Prevention criteria
* Children accompanied by the support center where the study was conducted.

Exclusion Criteria:

* Children who did not undergo assessments after the intervention
* Children those weighing < 9,600 kg, with uncontrolled seizures, or orthopedic changes (e.g., hip subluxations or dysplasia, severe spasticity combined with joint contractures, and severe scoliosis [Cobb angle > 40°]).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-88) | From enrollment to the end of treatment at 12 weeks
  This scale is widely used in children with neurological impairments, comprising 88 tasks divided into five dimensions: A (lying and rolling); B (sitting); C (crawling and kneeling); D (standing); and E (walking, running, and jumping). Each task received a score ranging from 0 (inability to start the task) to 3 (completes the task). Thus, the total GMFM-88 score ranged from 0 to 264 points; higher scores indicated better motor function.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Pesquisa Professor Joaquim Amorim Neto, Campina Grande, Paraíba, Brazil